CLINICAL TRIAL: NCT04956276
Title: A Phase 2, Multiple Ascending Dose, Randomized, Double-Blind, Placebo-Controlled Study of ALXN1830 Administered Subcutaneously in Patients With Warm Autoimmune Hemolytic Anemia (WAIHA)
Brief Title: Subcutaneous ALXN1830 in Adult Participants With Warm Autoimmune Hemolytic Anemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate program
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ALXN1830-WAI-202
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Warm Autoimmune Hemolytic Anemia
Keywords: Warm autoimmune hemolytic anemia; WAIHA; Immunoglobulin G-mediated autoimmune disorder; Pathogenesis; Anti-neonatal Fc receptor; ALXN1830
MeSH Terms: interventions — orilanolimab; rhoA GTP-Binding Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Cohorts 1 and 2 will be participant and investigator blinded, Cohort 3 will be open label (if initiated).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: ALXN1830/Placebo (Experimental): Participants will be randomized 3:1 to receive ALXN1830 or placebo. Treatment will be received for 8 weeks followed by a follow-up period (no treatment) for 8 weeks. Once complete, participants may continue participation in the study at the participant's and investigator's discretion during the OLE period for up to 2 years inclusive of primary treatment period.
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 2: ALXN1830/Placebo (Experimental): Participants will be randomized 3:1 to receive ALXN1830 or placebo. Treatment will be received for 8 weeks followed by a follow-up period (no treatment) for 8 weeks. Once complete, participants may continue participation in the study at the participant's and investigator's discretion during the OLE period for up to 2 years inclusive of primary treatment period.
  Interventions: Drug: ALXN1830; Drug: Placebo
- Cohort 3: ALXN1830 (Experimental): If initiated, participants will receive ALXN1830. Treatment will be received for 12 weeks followed by a follow-up period (no treatment) for 8 weeks. Once complete, participants may continue participation in the study at the participant's and investigator's discretion during the OLE period for up to 2 years inclusive of primary treatment period.
  Interventions: Drug: ALXN1830

INTERVENTIONS:
Drug: ALXN1830 — Administered as an SC infusion.
  Other Names: SYNT001 (formerly)
Drug: Placebo — Administered as an SC infusion.
  Arms: Cohort 1: ALXN1830/Placebo; Cohort 2: ALXN1830/Placebo

SUMMARY:
This is a Phase 2, multiple ascending, dose-finding, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, health-related quality of life, tolerability, pharmacokinetic, pharmacodynamic, and immunogenicity, of up to 3 dose regimens of ALXN1830 administered subcutaneous(ly) (SC) in the treatment of WAIHA.

This study will include 2 randomized, double-blind, placebo-controlled cohorts (Cohorts 1 and 2) to evaluate an 8-week treatment regimen, and an optional third open-label cohort (Cohort 3) to evaluate an alternative 12-week dosing regimen. Participants may continue participation in this study at the participant's and investigator's discretion in an open-label extension (OLE) period, consisting of monthly visits to observe participants for relapse, which will require going back on active treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with primary or secondary WAIHA at least 6 weeks prior to Screening.
* Failed or have not tolerated at least one prior WAIHA treatment regimen, for example, corticosteroids, rituximab, azathioprine, cyclophosphamide, cyclosporine, mycophenolate mofetil, danazol, or vincristine.
* Hemoglobin < 10 g/dL and ≥ 6 g/dL at Screening.
* Positive direct antiglobulin test (Coombs) (IgG positive who are positive or negative for the presence of complement C3) at Screening.
* Evidence of active hemolysis including any one of the below:

  * LDH > upper limit of normal (ULN) or
  * Haptoglobin < lower limit of normal or
  * Indirect bilirubin > ULN
  * Total IgG > 500 mg/dL at Screening
  * Platelet count ≥ 75 x 10^9/liter (L)
  * Absolute neutrophil count greater than 1.0 x 10^9/L

Key Exclusion Criteria:

* Participants with Evan's syndrome.
* Human immunodeficiency virus (HIV) infection (positive HIV 1 or HIV 2 antibody test).
* Positive hepatitis B surface antigen or hepatitis C antibody test.
* Inability to travel to the clinic for specified visits during the Primary Treatment Period or fulfill the logistical requirements of study intervention administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion Of Participants Achieving A ≥ 2 Grams/Deciliter (g/dL) Increase In Hemoglobin (Hgb) From Baseline To The End Of Primary Treatment | Baseline through Week 12
  Participants will have to achieve this increase without requiring any increase in the dose of an existing WAIHA medication after Day 1 (baseline) and without packed red blood cells (pRBC) transfusions after Day 14.

SECONDARY OUTCOMES:
Total Number Of Units Of pRBCs Transfused | Baseline through Week 12
Number Of Hgb Measurements ≥ 2 g/dL From Baseline To The End Of Primary Treatment | Baseline, Week 12
Time To Hgb Increase By ≥ 2 g/dL From Baseline | Baseline through Week 12
Proportion Of Participants Who Require New WAIHA Rescue Medication Or Any Increase In The Dose Of An Existing WAIHA Medication Or pRBC Transfusions For The Treatment Of Anemia | Day 15 through Week 12
Proportion Of Participants Achieving A ≥ 2 g/dL Increase In Hgb From Baseline Through Week 4 | Baseline through Week 4
  Participants need to achieve this increase without requiring any increase in the dose of an existing WAIHA medication after Day 1 and without pRBC transfusions after Day 14.
Change From Baseline To The End Of Primary Treatment In Serum Lactate Dehydrogenase (LDH) Levels | Baseline, Week 12
Change From Baseline To The End Of Primary Treatment In Absolute Reticulocyte Count | Baseline, Week 12
Change From Baseline To The End Of Primary Treatment In Serum Indirect Bilirubin | Baseline, Week 12
Change From Baseline To The End Of Primary Treatment In Serum Haptoglobin | Baseline, Week 12
Total Corticosteroid Usage From Baseline To The End Of Primary Treatment | Baseline, Week 12
Proportion Of Participants Who Require Any Increase In Corticosteroid Dose From Baseline To The End Of Follow Up After Primary Treatment | Baseline through Week 20
Change In Corticosteroid Dose From The End Of Primary Treatment To The End Of Follow Up | Week 12, Week 20
Number Of Days To Beginning Of Corticosteroid Taper During Follow Up After Primary Treatment | Baseline through Week 20
  Taper is defined as the first day that a lower dose of corticosteroids is prescribed/taken.
Number Of Days To Corticosteroid Maintenance Dose During Follow Up After Primary Treatment | Baseline through Week 20
  Maintenance dose will be defined as < 10 milligrams (mg)/day of prednisone or equivalent.
Number Of Days To Reach Corticosteroid Discontinuation From The End Of Primary Treatment To The End Of Follow Up After Primary Treatment | Week 12 through Week 20
Incidence And Titers Of Anti-drug Antibodies Against ALXN1830 Over Time | Up to 2 years
Incidence And Titers Of Neutralizing Antibodies Against ALXN1830 Over Time | Up to 2 years
Serum Trough Concentrations Of ALXN1830 Over Time | Up to 2 years
Change In Serum Total Immunoglobulin G (IgG) Levels By Dose Group And Time Point | Up to 2 years
Change From Baseline Of IgG Subtypes (IgG1 4) By Dose Group And Time Point | Up to 2 years
Change From Baseline Of IgA By Dose Group And Time Point | Up to 2 years
Change From Baseline Of IgM By Dose Group And Time Point | Up to 2 years
Change From Baseline Of Albumin By Dose Group And Time Point | Up to 2 years
Change From Baseline Of Circulating Immune Complexes By Dose Group And Time Point | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Study Site, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Yes